CLINICAL TRIAL: NCT00288808
Title: Comparison Between Point of Care Device and Venous Blood International Normalized Ratio Measurements for Pediatric Patients on Anticoagulation Therapy.
Brief Title: Comparison Between Point of Care Device and Venous Blood International Normalized Ratio Measurements.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: insufficient enrollment
Sponsor: University of Rochester (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 11787
Record Dates: First submitted 2006-02-06; First posted 2006-02-08 (Estimated); Last update posted 2015-04-27 (Estimated); Status verified 2015-04

CONDITIONS: Blood Coagulation Disorder
Keywords: Blood; Coagulation; PT/InR; Warfarin; Mechanical Valve
MeSH Terms: conditions — Blood Coagulation Disorders; Thrombosis

INTERVENTIONS:
Device: Hemosense (PT/InR point of care device)

SUMMARY:
Investigate the validity of Hemosense System in pediatric patients on anticoagulation therapy.

DETAILED DESCRIPTION:
Over the last few decades there has been an increased use of Warfarin in the pediatric population stemming from the use of mechanical heart valves and palliative surgical procedures requiring anticoagulation therapy. Other patients with enzymatic deficiency within the coagulation cascade may develop thrombosis treated with anticoagulation, i.e. factor V Leiden deficiency. Prevention of poor outcome from thrombosis has required closer monitoring in the pediatric patient. In addition, absorption of Warfarin in the pediatric population is highly variable and depends on the child's age, weight, diet, and concurrent use of other medications (Desai, 2000). This makes achieving anticoagulation very difficult. "Because of the intrinsic differences in the coagulation systems in children and adults, guidelines for antithrombotic therapy in adults cannot be extrapolated to pediatrics" (Desai, 2000). Therefore, pediatric patients on anticoagulation therapy require frequent lab work to monitor their prothrombin time and international ratios (PT/INR).

There are a number of barriers to care when discussing anticoagulation therapy for pediatric patients. Frequent venous blood draws represent a painful procedure that elicit anxiety and fear which leads to noncompliance. In addition, children are more difficult to obtain blood samples because of smaller vessels, patient movement during procedure, and the volume of blood that is required for the test. Other barriers include the time delay from when the patient has the lab work drawn, to when the result get to the provider for any patient care decisions to be made.

There are a number of Point of Care devices available for near-patient testing of the PT/InR's that requires only a finger stick. These monitors have been validated against standardized laboratory testing, in order for the monitor to be certified by the FDA. Similar studies to validate finger stick methods in pediatric patients have not been completed. The aim of this project is to validate the accuracy of Hemosense, a point of care device, to venous blood PT/InR level in the pediatric population.

ELIGIBILITY:
Inclusion Criteria:

- All pediatric patient requiring Warfarin therapy.

Exclusion Criteria:

1. Subjects older then 18 year of age.
2. Pregnant subjects.

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2005-10; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
The compariative accuracy between Point of Care device and standard of care method of determining PT/InR (Laboratory testing using Venous blood Draw)

CONTACTS AND LOCATIONS:
Overall Officials: Peter H Chang, D.O., Principal Investigator — University of Rochester Strong Memorial Hospital
Locations (1):
- University of Rochester Strong Medical Center, Rochester, New York, United States

REFERENCES:
- [Background] Poller L, Keown M, Chauhan N, van den Besselaar AM, Meeuwisse-Braun J, Tripodi A, Clerici M, Jespersen J. European concerted action on anticoagulation. Use of plasma samples to derive international sensitivity index for whole-blood prothrombin time monitors. Clin Chem. 2002 Feb;48(2):255-60. PMID 11805005